CLINICAL TRIAL: NCT02699983
Title: Virtual Weight Loss Program for African-American Breast Cancer Survivors
Brief Title: eHealth Weight Loss Program in African American Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeanne M. Ferrante, MD, MPH, Professor, Deparment of Family Medicine, RWJMS, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro20150001595; NCI-2015-02137 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20150001595 (Other: Rutgers University eIRB); 131404 (Other: Rutgers Cancer Institute of New Jersey); R21CA191431 (NIH)
Record Dates: First submitted 2016-03-01; First posted 2016-03-07 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Cancer Survivor; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage 0 Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ | interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (SparkPeople program) (Experimental): Participants receive one 30-minute session with the research assistant for training on how to use the SparkPeople website, and they may request additional training if needed.
  Participants are instructed to self-monitor their diet at least weekly using the SparkPeople tool, and to self-monitor their activity daily using the Fitbit monitoring device.
  Participants receive weekly motivational reminders to log into the website for 3 months via email, text, or phone, based on patient preference (active phase). Participants then enter the maintenance phase for 3 months without reminders.
  All participants answer survey questions on quality of life and social cognitive theory variables and undergo anthropometric measurements at baseline, 3, and 6 months.
  Interventions: Behavioral: Behavioral Dietary Intervention; Behavioral: Exercise Intervention; Device: Activity Monitoring Device
- Group II (wait list) (Active Comparator): Participants receive the weight loss handout and a Fitbit activity monitoring device and proceed with their usual life. After 6 months, patients receive the SparkPeople treatment as in Group I. All participants answer survey questions on quality of life and social cognitive theory variables and undergo anthropometric measurements at baseline, 3 and 6 months.
  Interventions: Device: Activity Monitoring Device

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Use SparkPeople web-based program
  Arms: Group I (SparkPeople program)
Behavioral: Exercise Intervention — Use Fitbit monitor and SparkPeople web-based program
  Arms: Group I (SparkPeople program)
Device: Activity Monitoring Device — Wear Fitbit activity monitoring device
  Other Names: Monitor

SUMMARY:
This randomized pilot clinical trial studies how well a virtual weight loss program (SparkPeople) works in helping female African American breast cancer survivors maintain a healthy weight. Many patients with breast cancer are overweight or gain weight after diagnosis. SparkPeople is a free web-based weight loss program that features educational and motivational articles and videos, self-monitoring tools, incentives, social support communities (including discussion forums, teams, challenges, and expert blogs), and options for content to be delivered to members' email. It is a comprehensive program that includes advice on diet, physical activity, and behavioral strategies (such as self-monitoring diet and exercise), and emphasizes safe weight loss and receiving medical attention regularly when needed. A web-based program such as SparkPeople may help breast cancer survivors maintain a healthy weight, which may reduce the risk of cancer returning and patient fatigue, and improve patient quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine feasibility of using a free online commercial weight loss program (SparkPeople) in African-American (AA) breast cancer survivors, as measured by: 1) Accrual: percent (%) patients recruited and completing baseline assessments; 2) Study retention: % patients completing 6 month follow-up assessment; 3) Intervention adherence and sustainability (measured at 3, 6, 12 months): a) use of website- number of log-ins, time spent, and use of features such as food diaries, joining teams, posting on message boards (provided by SparkPeople); b) use of Fitbit monitor- % patients who wore the monitor and synced data; c) satisfaction (e.g., ease of use of website, usefulness of content, extra training and support needed) and barriers to participation (e.g., lack of computer access, lack of skills, time, interest, etc.).

SECONDARY OBJECTIVES:

I. Collect preliminary data on effect sizes of changes in our outcomes and potential mediators associated with the use of the online weight loss program.

OUTLINE: Patients are randomized to 1 of 2 groups.

All patients receive a handout of their personalized goals for weight loss, diet, and physical activity, with instructions to proceed slowly and as tolerated. Patients also wear a Fitbit monitoring device to monitor physical activity levels daily.

GROUP I: Patients receive one 30-minute session with the research assistant for training on how to use the SparkPeople website, and may request additional training if needed. Patients are instructed to self-monitor their diet at least weekly using SparkPeople and physical activity levels daily using the Fitbit monitoring device, which integrates with the SparkPeople program. Patients receive weekly motivational reminders to log into the website for 3 months via email, text, or phone, based on patient preference (active phase). Patients then enter the maintenance phase for an additional 3 months without reminders.

GROUP II: Patients receive the weight loss handout and a Fitbit health monitoring device and proceed with their usual life. After 6 months, patients receive the SparkPeople treatment as in Group I.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have evidence of histologically confirmed breast cancer, stage 0, I, II or III, and be at least 2 years post diagnosis
* Patient is self-identified as African-American
* Patient is overweight or obese (body mass index [BMI] >= 25 kg/m^2)
* Patient is able to understand and read English
* Patient must have home internet or smartphone access
* Patient must give informed consent for this new study

Exclusion Criteria:

* Patient has a serious medical condition (e.g., stroke, liver or renal failure, congestive heart failure, myocardial infarction or cardiac surgery in past year, angina pectoris) that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator
* Patient has serious psychiatric condition (e.g., bipolar disorder, schizophrenia or other psychosis, bulimia or anorexia nervosa, suicide attempt within 6 months or current active suicidal ideation) that would compromise the patient's ability to complete the study, at the discretion of the investigator
* Patient has severe disabilities limiting moderate physical activity, such as severe orthopedic conditions
* Patient is planning major surgery within the next 6 months
* Patient is taking medications or supplements for weight loss currently or within the past 3 months
* Patient has successfully lost 5% of body weight in the previous 6 months or has had bariatric surgery
* Patient is pregnant, breastfeeding, has given birth within the last 3 months or planning pregnancy within the next 12 months; if participant becomes pregnant during the course of the study, she will be removed from further participation
* Patient is anticipating leaving the area within the next 12 months

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Ferrante, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

REFERENCES:
- [Derived] Ferrante JM, Devine KA, Bator A, Rodgers A, Ohman-Strickland PA, Bandera EV, Hwang KO. Feasibility and potential efficacy of commercial mHealth/eHealth tools for weight loss in African American breast cancer survivors: pilot randomized controlled trial. Transl Behav Med. 2020 Oct 8;10(4):938-948. doi: 10.1093/tbm/iby124. PMID 30535101

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I (SparkPeople Program): Participants receive training on how to use the SparkPeople website, self-monitor their diet using the SparkPeople tool, and to self-monitor their activity daily using the Fitbit monitoring device.
  Participants receive weekly motivational reminders to log into the website for 3 months via email, text, or phone, based on patient preference (active phase). Participants then enter the maintenance phase for 3 months without reminders.
  Behavioral Dietary Intervention: Use SparkPeople web-based program
  Exercise Intervention: Use Fitbit monitor and SparkPeople web-based program
  Activity Monitoring Device: Wear Fitbit activity monitoring device
- Group II (Wait List): Participants receive the weight loss handout and a Fitbit activity monitoring device and proceed with their usual life. After 6 months, patients receive the SparkPeople treatment as in Group I.
  Activity Monitoring Device: Wear Fitbit activity monitoring device
Period: Overall Study
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Started | 18 | 17
Completed | 17 | 17
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group II (Wait List): Participants receive the weight loss handout and a Fitbit activity monitoring device and proceed with their usual life. After 6 months, patients receive the SparkPeople treatment as in Group I.
- Total: Total of all reporting groups
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List) | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.20 (10.26) | 62.25 (6.66) | 61.67 (8.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 14 | 17 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 17 | 35
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35
BMI [Mean (Standard Deviation); unit: kg/m^2] | 35.51 (6.98) | 38.40 (6.94) | 36.73 (6.84)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: Number of eligible participants who were enrolled and randomly assigned. Feasibility is defined as >= 75% recruitment rate.
Time Frame: 12 months
Population: The overall number of participants is the number that were eligible for the study, hence it is greater than the number with results.
Measure: Count of Participants; unit: Participants
Groups:
- Group II (Wait List): Participants receive the weight loss handout and a Fitbit activity monitor. After 6 months, participants receive the SparkPeople treatment.
  Exercise Intervention: Use Fitbit monitor
  Activity Monitoring Device: Wear Fitbit activity monitoring device
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 23 | 22
Participants | 18 | 17

2. Primary Outcome: Retention Rate
Description: Number of participants completing study. Feasibility will be defined as >= 80% retention rate.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Group II (Wait List): Participants receive a weight loss handout and a Fitbit activity monitoring device and proceed with their usual life. After 6 months, patients receive the SparkPeople treatment as in Group I.
  Exercise Intervention: Use Fitbit monitor
  Activity Monitoring Device: Wear Fitbit activity monitoring device
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
Participants | 17 | 17

3. Primary Outcome: Adherence to SparkPeople- Logged in
Description: average number of days logged per week in to SparkPeople website
Time Frame: 0-3 months after intervention
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
days/week | 3.01 (2.07) | 2.30 (2.27)

4. Primary Outcome: Adherence to SparkPeople- Logged in
Description: Average number of days per week logged in to SparkPeople website
Time Frame: 4-6 months after intervention
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
days/week | 2.30 (2.30) | 1.14 (1.64)

5. Primary Outcome: Adherence to SparkPeople- Logged Food
Description: Average number of days per week logged food into SparkPeople
Time Frame: 0-3 months after intervention
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
days/week | 1.69 (1.84) | 1.50 (1.85)

6. Primary Outcome: Adherence to SparkPeople- Logged Food
Description: Average number of days per week logged food into SparkPeople
Time Frame: 4-6 months after intervention
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
days/week | 0.6 (0.87) | 0.71 (1.17)

7. Primary Outcome: Acceptability of SparkPeople
Description: Usefulness of SparkPeople website on 1 (not useful at all) to 4 (very useful) scale
Time Frame: 0-3 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
score on a scale | 3.53 (0.83) | 3.60 (0.52)

8. Primary Outcome: Acceptability of SparkPeople
Description: Usefulness of SparkPeople website on 1 (not useful at all) to 4 (very useful) scale
Time Frame: 4-6 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
score on a scale | 3.53 (0.80) | 3.42 (0.79)

9. Primary Outcome: Adherence to Fitbit
Description: average days used Fitbit per week
Time Frame: 0-3 months after intervention
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
days/week | 6.24 (0.84) | 5.96 (1.63)

10. Primary Outcome: Adherence to Fitbit
Description: average days used Fitbit per week
Time Frame: 4-6 months after intervention
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
days/week | 5.57 (1.83) | 5.61 (1.77)

11. Primary Outcome: Acceptability of Fitbit
Description: Usefulness of Fitbit, rated on 1 (not useful at all) to 4 (very useful) scale
Time Frame: 0-3 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
score on a scale | 3.93 (0.26) | 3.93 (0.26)

12. Primary Outcome: Acceptability of Fitbit
Description: Usefulness of Fitbit, rated on 1 (not useful at all) to 4 (very useful) scale
Time Frame: 4-6 months after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
score on a scale | 4.00 (0) | 4.00 (0)

13. Secondary Outcome: Change in Weight
Description: Change in weight from baseline
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
kg | -2.10 (2.64) | -2.26 (2.16)

14. Secondary Outcome: Change in Weight
Description: Change in weight from baseline
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
kg | -1.71 (1.88) | -2.53 (4.00)

15. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
cm | -1.98 (5.39) | -0.05 (5.56)

16. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
cm | -3.56 (4.70) | -0.84 (5.21)

17. Secondary Outcome: Change in Caloric Intake
Description: Changes in caloric intake per day, measured by 24-hour recall
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
kcal/day | -62.06 (589.27) | -386.38 (514.95)

18. Secondary Outcome: Change in Caloric Intake
Description: Changes in caloric intake per day, measured by 24-hour recall
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
kcal/day | -216.65 (606.09) | -173.06 (805.40)

19. Secondary Outcome: Change in Physical Activity
Description: change in average number of steps per day measured using Fitbit monitor
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
steps per day | 466.36 (2203.49) | -609.83 (2898.36)

20. Secondary Outcome: Change in Physical Activity
Description: change in average number of steps per day measured using Fitbit monitor
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
steps per day | -107.07 (2184.94) | -205.47 (2147.79)

21. Secondary Outcome: Cardiopulmonary Fitness
Description: change in fitness, measured by the 6-minute walk test
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
meters | 0.81 (51.13) | 20.07 (52.81)

22. Secondary Outcome: Cardiopulmonary Fitness
Description: change in fitness, measured by the 6-minute walk test
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
meters | 26.64 (35.88) | 31.97 (26.27)

23. Secondary Outcome: Change in Quality of Life
Description: measured using Quality of Life in Adult Cancer Survivors Scale (minimum 65, maximum 257); higher scores mean worse quality of life
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
units on a scale | -5.44 (18.11) | -4.35 (16.69)

24. Secondary Outcome: Change in Quality of Life
Description: as for outcome 23
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
units on a scale | -9.44 (16.97) | -4.65 (24.21)

25. Secondary Outcome: Self-efficacy, Eating Healthy Foods
Description: change in self-efficacy, eating healthy foods, measured with Health Beliefs Survey, scale range 0 (certain I cannot) to 100 (certain I can)
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group I (SparkPeople Program): Participants receive training on how to use the SparkPeople website, self-monitor their diet using the SparkPeople tool, and to self-monitor their activity daily using the Fitbit monitoring device.
  Participants receive weekly motivational reminders to log into the website for 3 months via email, text, or phone, based on patient preference (active phase). Participants then enter the maintenance phase for 3 months without reminders.
  All participants have follow-up visits at 3, 6, 9, and 12 months to answer survey questions on quality of life and social cognitive theory variables and undergo anthropometric measurements.
- Group II (Wait List): Participants receive the weight loss handout and a Fitbit activity monitoring device and proceed with their usual life. After 6 months, patients receive the SparkPeople treatment as in Group I. All participants have follow-up visits at 3, 6, 9, and 12 months to answer survey questions on quality of life and social cognitive theory variables and undergo anthropometric measurements.
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
units on a scale | 2.14 (8.17) | -0.41 (13.47)

26. Secondary Outcome: Self-efficacy, Eating Healthy Foods
Description: as for outcome 25
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
units on a scale | 5.59 (12.63) | -6.59 (15.36)

27. Secondary Outcome: Social Support for Healthy Nutrition
Description: change in social support for healthy nutrition, measured by Health Beliefs Survey, scale range 1 (strongly disagree) to 5 (strongly agree); a higher number, e.g., 5 (strongly agree) is the more favorable outcome
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
units on a scale | 0.40 (0.58) | 0.11 (0.56)

28. Secondary Outcome: Social Support for Healthy Nutrition
Description: as for outcome 27
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
Number analyzed (Participants) | 18 | 17
units on a scale | 0.39 (0.85) | 0.11 (0.71)

ADVERSE EVENTS:
Time Frame: 6 months
Description: This is a minimal risk study. The lifestyle behavioral modification intervention did not place participants at risk for any serious adverse events or death.
Arm/Group | Group I (SparkPeople Program) | Group II (Wait List)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT02699983/Prot_SAP_000.pdf